CLINICAL TRIAL: NCT06284135
Title: Prospective Randomised Study to Examine the Influence of a Modification of the DaVinci Prostatectomy on the Frequency of Postoperative Lymphoceles Requiring Treatment and Postoperative Complications
Brief Title: MICHL-trial: Impact of Peritoneal Bladder Flap in RARP Patients on Lymphoceles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Martini-Klinik am UKE GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017-PS-03; PV6099 (Other: Martini-Klinik)
Record Dates: First submitted 2024-02-14; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Lymphocele After Surgical Procedure
Keywords: prostate cancer; radical prostatectomy; pelvic lymph node dissection; lymphocele; complication
MeSH Terms: conditions — Prostatic Neoplasms; Lymphocele

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Michl-stitch (Experimental)
  Interventions: Other: Michl-stitch
- control (No Intervention)

INTERVENTIONS:
Other: Michl-stitch — In the intervention group, a ventral fixation was performed by suturing the ventral bladder peritoneum to the plexus Santorini and from there to the right and left lateral endopelvic fascia (MICHL-stitch).
  Arms: Michl-stitch

SUMMARY:
A two-armed prospective randomised, controlled, single-centre trial on 1080 patients with prostate cancer who underwent robot-assisted radical prostatectomy with bilateral pelvic lymph node dissection was carried out. Patients in the intervention arm received fixation of the peritoneal flap of the bladder to the plexus Santorini at the end of surgery (Michl-technique, MT); in the control group, surgery was performed without this modification. The primary endpoint was the rate of lymphoceles requiring intervention.

ELIGIBILITY:
Inclusion Criteria:

* Declaration of consent signed
* Minimum age 18 years
* localised prostate carcinoma
* planned DVRP with bilateral lymphadenectomy

Exclusion Criteria:

* patient's lack of capacity to consent
* ORP
* no planned PLND
* metastatic prostate cancer
* ASA status >3

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1080 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
rate of lymphoceles requiring intervention after RARP | one year follow-up
  Clavien-Dindo >2°

SECONDARY OUTCOMES:
total lymphocele rate after RARP | one year follow-up
  Clavien-Dindo
other complications ≥ grade IIIa according to Clavien-Dindo after RARP | one year follow-up
  Clavien-Dindo
continence rates after RARP | one year folow-up
  EPIC

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Michl, Principal Investigator — Martini-Klinik am UKE GmbH
Locations (1):
- Martini-Klinik am UKE GmbH, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
A publication in a peer-reviewed journal is planned
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after final analysis
Access Criteria: peer-reviewed journal

REFERENCES:
- [Background] Ploussard G, Briganti A, de la Taille A, Haese A, Heidenreich A, Menon M, Sulser T, Tewari AK, Eastham JA. Pelvic lymph node dissection during robot-assisted radical prostatectomy: efficacy, limitations, and complications-a systematic review of the literature. Eur Urol. 2014 Jan;65(1):7-16. doi: 10.1016/j.eururo.2013.03.057. Epub 2013 Apr 6. PMID 23582879
- [Background] Keskin MS, Argun OB, Obek C, Tufek I, Tuna MB, Mourmouris P, Erdogan S, Kural AR. The incidence and sequela of lymphocele formation after robot-assisted extended pelvic lymph node dissection. BJU Int. 2016 Jul;118(1):127-31. doi: 10.1111/bju.13425. Epub 2016 Feb 17. PMID 26800257
- [Background] Waldert M, Remzi M, Klatte T, Klingler HC. FloSeal reduces the incidence of lymphoceles after lymphadenectomies in laparoscopic and robot-assisted extraperitoneal radical prostatectomy. J Endourol. 2011 Jun;25(6):969-73. doi: 10.1089/end.2010.0635. Epub 2011 May 4. PMID 21542773
- [Background] Yasumizu Y, Miyajima A, Maeda T, Takeda T, Hasegawa M, Kosaka T, Kikuchi E, Oya M. How can lymphocele development be prevented after laparoscopic radical prostatectomy? J Endourol. 2013 Apr;27(4):447-51. doi: 10.1089/end.2012.0356. Epub 2012 Dec 5. PMID 23030822
- [Background] Grande P, Di Pierro GB, Mordasini L, Ferrari M, Wurnschimmel C, Danuser H, Mattei A. Prospective Randomized Trial Comparing Titanium Clips to Bipolar Coagulation in Sealing Lymphatic Vessels During Pelvic Lymph Node Dissection at the Time of Robot-assisted Radical Prostatectomy. Eur Urol. 2017 Feb;71(2):155-158. doi: 10.1016/j.eururo.2016.08.006. Epub 2016 Aug 17. PMID 27544575
- [Background] Lebeis C, Canes D, Sorcini A, Moinzadeh A. Novel Technique Prevents Lymphoceles After Transperitoneal Robotic-assisted Pelvic Lymph Node Dissection: Peritoneal Flap Interposition. Urology. 2015 Jun;85(6):1505-9. doi: 10.1016/j.urology.2015.02.034. PMID 26099895